CLINICAL TRIAL: NCT00198198
Title: Open Label Pilot Study of Aripiprazole Treatment of Difficult to Treat Bipolar Depression
Brief Title: Aripiprazole Treatment of Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69883; 0402-46
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
This is a study of addition of aripirazole to the treatment of bipolar depressed patients who are not better on the medications that they are currently receiving.

DETAILED DESCRIPTION:
Hypothesis/Objectives:

Aim 1: To investigate whether aripiprazole is effective in the treatment of bipolar depression.

Hypothesis 1: Aripiprazole will lead to a significant decrease in scores on the Hamilton Depression Rating Scale (HAM-D) during an 8-week treatment course.

a. Study Population:

A total number of 10 evaluable patients will be enrolled in the study.

c. Study Design and Method

This proposal will use an open label design. Aripiprazole will be added to the treatment of patients with DSM-IV (American Psychiatric Association, 1994) BDD. Patients will be allowed to continue their psychotropic medication, at a stable dose, as long as they meet inclusion criteria as described below. Aripiprazole will be started at a dose of 10 mg for two weeks, 15 mg for an additional two weeks, and 20 mg for the last four weeks. The length of time a patient stays on the maximum dose (20 mg) depends upon the patient's tolerance and treatment response. Treatment will continue for 8 weeks with weekly visits and ratings on the 17-item Hamilton Depression Rating Scale (HAM-D 17) and other ratings scales.

ELIGIBILITY:
Inclusion Criteria:

* 1) Male or female between 18 - 65 years of age, inclusive 2) Satisfy DSM-IV criteria for bipolar disorder depressed phase i.e.,duration of depression > 2 weeks) 3) No change in psychotropic medication or their doses within 2 weeks of inclusion in The study. 4) Inadequately responsive to or intolerant of prior pharmacotherapy as determined by the investigator 5) 17-item Hamilton Depression Rating Scale Score > 15 6) Young Mania Rating Scale (Young, et. al., 1978) (YMRS) < 10.

Exclusion Criteria:

Exclusion Criteria: 1) History of or currently suffering from serious medical illness, or be on medication that may interact with aripiprazole 2) On any other neuroleptic e.g., olanzapine, risperidone, ziprasidone, haloperidol.

3) History of substance abuse within 3 months or substance dependence within 6 months of the study. 4) Pregnant or planning to be pregnant or not using adequate contraception. 5) Received electroconvulsive therapy (ECT) treatment in the past 1 year. 6) Significant suicide or homicide risk at the time of the study; 7) Not on any herbal or any other alternative pharmacological treatment. 8) Renal or hepatic dysfunction 9) History of decreased sweating or heat stroke.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-08; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- UH 3124 University Hospital, Indianapolis, Indiana, United States